CLINICAL TRIAL: NCT06959433
Title: Safety and Efficacy of Lu-177 PSMA Treatment in Metastatic Clear Cell Renal Carcinoma
Brief Title: Lu-177 PSMA Treatment in Cell Renal Carcinoma
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Cigdem Soydal, Prof of Nuclear Medicine, Ankara University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Lu-PSMA RCC
Record Dates: First submitted 2025-04-28; First posted 2025-05-06 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-04

CONDITIONS: Metastatic Renal Cancer
Keywords: Renal Cell Carcinoma, Radionuclide treatment, efficacy, safety.
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — Pluvicto

STUDY DESIGN:
Intervention Model Description: a single arm will be included patients with metastatic RCC treated with Lu-177 PSMA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lu-PSMA treatment arm (Experimental): Patients who will received Lu-177 PSMA treatment for metastatic RCC
  Interventions: Drug: Lu-177 PSMA-617

INTERVENTIONS:
Drug: Lu-177 PSMA-617 — Included patients will receive 4 cycles of 7.4GBq Lu-177 PSMa therapy every 6 weeks. If any toxicity develops after the first cycle, dose reduction will be performed for the other cycles. At 1. And 4. Cycles of therapy, whole body planar and SPECT/CT imaging will be performed at 4. And 24. Hours and any time at 4-7.days of injection. On these images , kindey, liver and salivary gland doses will be calculated. Mean tumor dose will also be calculated by measurinf the tumoral uptake. In the follow up, patients will be controlled at 9. And 24. Weeks and every 12 months then after.

SUMMARY:
Summary Renal Cell Carcinoma (RCC) consists of 2% of all malignencies. RCCs are generally divided to histopathological subtypes as clear cell and non-clear cell variants. Clear cell variant responsible for the 75-80% of all RCCs. It is reported that 20-30% of RCCs are metastatic at the diagnosis and 5 years survival is approximately is 10-20% in this group of patients. Moreover, 60% of patients who are not metastatic at the diagnosis, develop metastates within 2-3 years. 2nd and 3th line effective treatment option in metastatic RCCs patients has been a subject of interest.

PSMA (protatate specific membrane antigen) with the other name glutamate carboxypeptidase, is a transmembrane protein and overexpresses in prostate adenocarcinomas and neoangiogenesis spots of endothelium of other several tumor types. It infronts as a target for theranostic consept for mainly prostate cancer in nuclear medicine. As a radionuclide treatment option, Lu-177 PSMA treatment is proved as safe and effective treatment option in castration resistant prostata cancer patients. After its widely use in prostate cancer, it is reported that PSMA molecule can be used for imaging of RCC patients and PSMA uptake is higher than 18F-FDG. For this reason, Lu-177 PSMA treatment can be a systemic treatment option in RCC patients who have progress afer 1st cycle treatment. In this study we aimed to safety and efficacy of Lu-177 PSMA treatment in metastatic RCC patients as systemic radionuclide treatment option.

ELIGIBILITY:
Inclusion Criteria:

* Age >18
* Progression after at least 2 lines of systemic therapy or existence of a contraindication to systemic therapies
* At least 3 years of life expectancy
* ECOG performance status ≤ 2
* Ability to sign informed consent

Exclusion Criteria:

* Age<18
* Not having received any systemic therapies
* History of a secondary malignancy
* ECOG performance status > 2
* Any contraindication for radionuclide therapy (pregnancy, lactation, organ disfunction, metastatic lesions with a risk of compression
* Previous history of any radionuclide therapies
* Inability to sign informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2028-02-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
toxicity analysis | 1-36 months
  Therapy associated toxicity will be evaluated according to CTCAE V5.0 criteria.

SECONDARY OUTCOMES:
efficacy analysis | 1-36 months
  Therapy response will be evaluated according to RECIST 1.1 criteria

IPD SHARING:
Plan to Share IPD: Undecided